CLINICAL TRIAL: NCT03259594
Title: Measurement of Renal Functional Reserve Change In Patients With Simple Renal Cysts Before and After Laparoscopic Deroofing
Brief Title: Measurement of Renal Functional Reserve Change In Patients With SRC Before and After Laparoscopic Deroofing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ou tongwen (Other)
Responsible Party: Sponsor-Investigator, ou tongwen, Head of Urology, Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: otw-20170804-01
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Simple Renal Cyst
Keywords: Renal functional reserve; Simple renal cysts; Laparoscopic deroofing

STUDY DESIGN:
Intervention Model Description: Participants are assigned to two groups.One group participants are with endophytic simple renal cysts, and the other are with exophytic simple renal cysts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endophytic group (Experimental): participants are with endophytic renal cyst and undergo laparoscopic deroofing.2 day before laparoscopic deroofing, they were given intravenous 100 g of amino acids supplementation.
  Interventions: Procedure: Laparoscopic deroofing; Drug: 100 g of amino acids supplementation
- exophytic group (Sham Comparator): participants are with exophytic renal cyst and undergo laparoscopic deroofing.2 day before laparoscopic deroofing, they were given intravenous 100 g of amino acids supplementation.
  Interventions: Procedure: Laparoscopic deroofing; Drug: 100 g of amino acids supplementation

INTERVENTIONS:
Procedure: Laparoscopic deroofing — The classic treatment of patients with simple renal cysts is deroofing, which can be performed by open surgery or laparoscopy. Laparoscopic deroofing is an effective minimally invasive approach and has gained popularity.
Drug: 100 g of amino acids supplementation — intravenous supplementation with 100 g of amino acids 2 day before laparoscopic deroofing.
  Other Names: Compound Amino Acids Injection(18AA-Ⅶ)

SUMMARY:
Renal functional reserve may be improved in patients with simple renal cysts after laparoscopic deroofing.

DETAILED DESCRIPTION:
Simple renal cysts (SRC) are the most frequent type of cystic renal disease. The prevalence rate of SRCs is about 10% and increases with age. Hypertension and decreased renal functions have been reported to occur more commonly among these patients with SRC and there are no clear guidelines for managing asymptomatic SRCs.Renal functional reserve (RFR) describes the capacity of the intact nephron mass to increase glomerular filtration rate(GFR) from baseline in response to stimuli (e.g., protein load).The investigators hypothesized that RFR may be improved in some patients with simple renal cysts after laparoscopic deroofing despite identical resting glomerular filtration rate (rGFR).The aim of this study is to examine whether there is improvement of RFR in patients with simple renal cysts after laparoscopic deroofing.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18
2. Estimated GFR >30 mL/min/1.73m2
3. Subjects who signed informed consent forms

Exclusion Criteria:

1. Allergy to iothalamate, shellfish or iodine
2. Use of metformin or amiodarone
3. Inability to maintain a stable regimen of medications which affect GFR for > one week prior to participation (e.g. non-steroidal anti-inflammatory drugs, angiotensin converting enzyme inhibitors, angiotensin receptor blockers)
4. Use of medications which directly affect elimination of creatinine (e.g. cimetidine and trimethoprim)
5. Acute exacerbation of asthma or chronic obstructive pulmonary disease within 3 months requiring hospitalization or oral steroid therapy
6. Inadequate intravenous access
7. Severe anemia (Hct <21%)
8. Acute kidney injury (rise in creatinine to ≥1.5 times the previous baseline or by ≥ 0.3 mg/dL on most recent labs prior to enrollment)
9. History of contrast-induced nephropathy
10. Hyperthyroidism
11. Pheochromocytoma
12. Sickle cell disease
13. Urinary retention or incontinence
14. Status post organ transplant
15. Pregnancy or active breast feeding
16. Cognitive impairment with inability to give consent
17. Institutionalized status

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in renal functional reserve after laparoscopic deroofing | 1 month after surgery.
  1 month after surgery, repeated glomerular filtration rate measurements are to be performed to calculate change in renal functional reserve.

CONTACTS AND LOCATIONS:
Overall Officials: Tongwen Ou, MD., Study Chair — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No